CLINICAL TRIAL: NCT06192043
Title: Cognitive Behavioral Interventions for Motivation, Psychological Distress and Quality of Life Among Individuals With Smoking Cessation: A Randomized Control Trial
Acronym: CBIMPDQLISC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Government College University Faisalabad (Other)
Responsible Party: Principal Investigator, Qasir Abbas, Dr. Qaisir Abbas Assisstant Professor Clinical Psychology, Government College University Faisalabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Govt.GCUF
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Cognitive Behavior Intervention for Psychological Distress, Motivation and Quality of Life Among Individual With Smoking Cessation
Keywords: Psychological Distress, Quality of Life, Motivation, Cognitive Behavior Therapy, Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Intervention Model Description: Randomized Control trial would be used in this study. It would be two two-arm study and two groups: The experimental and the control group. The experimental group will receive an intervention waitlist. In this research, a parallel group design will be used. We will give treatment to all participants in a parallel way. The allocation ratio and framework would be equivalence i.e., the treatment group and control group would be an equal number of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental treatment group (Experimental): Experimental Group:
  Participants in the experimental group would receive 6-8 sessions of Psychoeducational based program
  Waitlist Control group:
  Participants in the control group would not receive a psychoeducational-based Program
  Interventions: Behavioral: Behavioral Psychoeducational Intervention
- No intervention Control Group (No Intervention): Control Group:
  Participants in the control group didn't receive any Psychoeducational Intervention or any treatment

INTERVENTIONS:
Behavioral: Behavioral Psychoeducational Intervention — Psychoeducational Program would be used as an intervention strategy for individuals with smoking cessation to provide understanding and insight to the participants about the problem. Furthermore, this program would deal with interventions like motivation, cognitive conceptualization, coping skills and training, craving management, and relapse prevention among individuals with smoking cessation
  Arms: Experimental treatment group

SUMMARY:
The main purpose of this research is to find out how brief cognitive behavior intervention influences the motivation level, psychological distress, and quality of life among people with smoking cessation. Another objective of this research is to examine the effectiveness of cognitive behavioral therapy (CBT) among smoking people, another objective of this study is to investigate how Cognitive behavioral therapy helps to enhance the motivation level and quality of life and minimize psychological distress among people with smoking cessation

DETAILED DESCRIPTION:
Participants:

This was basically pre and post study, initially 60 sixty research participants were recruited for pre-assessment, while 4 participants left due to some reasons (2 persons went out of the city for a job, 1 person met a severe road accident, and 1 person simply refused to participate in this study furthermore. Finally, 55 research participants were recruited for post-assessment. These research participants belong to different residential areas (rural/urban) have varied family systems (nuclear/joint) have different birth order, education, socioeconomic status, education, occupation, marital status, and distant smoking duration. The data were analyzed with the help of SPSS-23 (Statistical Package for Social Sciences - 23) descriptive statistics, correlation analysis, and repeated measure ANOVA were used to understand the association and differences among pre and post-assessment of smoking personals.

ELIGIBILITY:
Inclusion Criteria:

* If we talk about inclusion criteria, the individuals who were ready to change their lives were part of this study, furthermore, persons above 18 years and below 60 years old were recruited for this study, minimum duration for smoking personnel was not less than 6 months and not more than 5 years were part of this study. The individuals who have signed a written informed consent form were part of this study. Moreover, only males who were easily comprehended and understood the instructions of the researcher were recruited in this study. On the other hand, if we talk about the exclusion criteria of the study

Exclusion Criteria:

* the individuals who were reluctant to participate, or had any kind of psychophysiological illness prior to the study were excluded from this research. Further, the people below 18 and above 60 years were excluded. Furthermore, the research participants who had any kind of trauma during this study were excluded and those who refused to become further part of this study were excluded from this research study.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-04-10 (Estimated)

PRIMARY OUTCOMES:
Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) | 6 months
  The ASSIST (Alcohol, Smoking and Substance Involvement Screening Test) was developed under the supervision of WHO (World Health Organization) by a group of researchers, clinicians, public health providers in 2010 (WHO, 2010). It mainly screens out the individual tendency to use Alcohol, Tabaco and other substances. This test mainly has seven items, which shows good test-retest reliability ranging from 0.6 to 0.8 (Humeniuk, 2008).
Cigarette Dependency scale (CDS) | 6 months
  The CDS (Cigarette Dependency scale) was developed by Jean-Francois Etter, PhD in 2003. (CDS; Etter et al.,2023). This scale has twelve items which gauge the addiction level, smoking compulsion, tolerability and withdrawal tendency of a person.
Depression Anxiety Stress Scale (DASS) | 6 months
  The (DASS) Depression Anxiety Stress Scale was developed in the University of New South Wales Australia to assess the level of depression, anxiety and stress among students. The DASS-21 was developed by Lovibond and Lovibond in 1995 (Minh Thi Hong Le, 2017). In this study the Urdu translated version of DASS was used which were translated by Naeem and Kamal in 2018 (Naeem and Kamal, 2018). It is very reliable and valid tool to assess negative emotional state of depression, stress and anxiety. The overall reliability of DASS is 0.74.
Motivation and Attitude towards changing Health (MATCH) | 6 months
  The MATCH (Motivation and Attitude towards changing Health) was developed by Hessler, Fisher, Polonsky, Browyer and Potter in 2018 (Hessler DM, Fisher L, Polonsky WH, Browyer V & Potter M., 2018). It's basically consist 9 items with 5 points Likert's scale ranging from strongly disagree to strongly agree).

CONTACTS AND LOCATIONS:
Overall Officials: Qasir Abbas, PHD, Principal Investigator — Government College University Faisalabad
Locations (1):
- GCUF, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No